CLINICAL TRIAL: NCT02642042
Title: A Phase II Trial of Trametinib With Docetaxel in Patients With KRAS Mutation Positive Non-Small Cell Lung Cancer (NSCLC) and Progressive Disease Following One or Two Prior Systemic Therapies
Brief Title: Trametinib and Docetaxel in Treating Patients With Recurrent or Stage IV KRAS Mutation Positive Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-02250; NCI-2015-02250 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1507; S1507 (Other: SWOG); S1507 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2015-12-29; First posted 2015-12-30 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: KRAS Gene Mutation; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; trametinib; omipalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (trametinib, docetaxel) (Experimental): Patients receive trametinib PO on days 1-21. Patients also receive docetaxel IV on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Trametinib

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK 212; GSK-1120212; GSK-212; GSK1120212; GSK212; JTP 74057; JTP-74057; JTP74057; MEK Inhibitor GSK1120212

SUMMARY:
This phase II trial studies how well trametinib and docetaxel work in treating patients with stage IV KRAS mutation positive non-small cell lung cancer or cancer that has come back. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving trametinib with docetaxel may work better in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate (confirmed and unconfirmed) to trametinib plus docetaxel in the entire study population of Kirsten rat sarcoma viral oncogene homolog (KRAS) mutation positive non-small cell lung cancer (NSCLC) patients following one or two prior systemic therapies.

SECONDARY OBJECTIVES:

I. To evaluate if trametinib plus docetaxel is consistent with promise of activity measured by the response rate in G12C KRAS mutation positive NSCLC patients following one or two prior systemic therapies.

II. To assess the response rate of this combination in non-G12C KRAS mutation positive NSCLC patients.

III. To assess progression-free survival within the G12C and non-G12C KRAS positive subgroups and the entire study population.

IV. To evaluate the toxicity of the regimen. V. To assess overall survival within G12C positive patients, non-G12C positive patients, and the entire study population.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To evaluate the response rates in the presence of comutations p53 and LKB1. II. To bank specimens for future research.

OUTLINE:

Patients receive trametinib orally (PO) on days 1-21. Patients also receive docetaxel intravenously (IV) on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* DISEASE RELATED CRITERIA: Patients must have pathologically confirmed KRAS mutation (at codon 12, 13 and 61) positive non-small cell lung cancer (NSCLC) that is stage IV or recurrent; the specific subtype of KRAS mutation must be known; KRAS mutation testing must have been performed in a Clinical Laboratory Improvement Act (CLIA) certified laboratory; CLIA certified commercially available tests are acceptable
* DISEASE RELATED CRITERIA: Patients must have measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI) within 28 days prior to registration; the CT from a combined positron emission tomography (PET)/CT may be used only if it is of diagnostic quality; non-measurable disease must be assessed within 42 days prior to registration; all known sites of disease must be assessed and documented on the baseline tumor assessment form (Response Evaluation Criteria in Solid Tumors [RECIST 1.1])
* DISEASE RELATED CRITERIA: Patients must not have known brain metastases, leptomeningeal carcinomatosis or spinal cord compression unless: (1) metastases have been locally treated (including stereotactic body radiation therapy [SBRT], whole brain radiotherapy [WBRT], and surgical resection) and have remained clinically controlled and asymptomatic for at least 14 days following treatment and prior to registration, AND (2) patient has no residual neurological dysfunction and has been off corticosteroids for at least 2 days prior to registration
* PRIOR/CONCURRENT THERAPY CRITERIA: Patients must have documented progressive cancer following at least one but no more than two prior regimens of systemic therapy for lung cancer, one of which must have been platinum based combination chemotherapy; treatment with an immune therapy or targeted therapy for advanced disease will be considered a separate regimen and will count toward the prior regimens; maintenance therapy will not be counted as a separate regimen; adjuvant chemotherapy or chemotherapy administered as part of concurrent chemotherapy and radiation therapy for the treatment of lung cancer will not count as a prior regimen of systemic therapy as long as recurrence of patient's lung cancer occurred more than 12 months after the last day of chemotherapy
* PRIOR/CONCURRENT THERAPY CRITERIA: Patients must not have received any chemotherapy, biologic agent, or any investigational agent within 14 days prior to registration. Patients must have recovered from any adverse events to Common Terminology Criteria for Adverse Events (CTCAE) grade 0-1 prior to registration
* PRIOR/CONCURRENT THERAPY CRITERIA: Prior treatment with an anti-PD-1 or anti-PDL1 is not required
* PRIOR/CONCURRENT THERAPY CRITERIA: Patients must not have received prior docetaxel; patients must not have received therapy with a drug known to be either a mitogen-activated protein kinase (MEK) inhibitor or a phosphatidylinositol 3 kinase (PI3K)/v-akt murine thymoma viral oncogene homolog 1 (AKT)/mammalian target of rapamycin (mTOR) pathway inhibitor
* PRIOR/CONCURRENT THERAPY CRITERIA: Patients must have recovered from any adverse effects from prior therapy (except alopecia) to =< CTCAE grade 1 prior to registration
* PRIOR/CONCURRENT THERAPY CRITERIA: Patients may have had prior radiation therapy as long as it has not affected greater than 25% of the bone marrow and at least one measurable lesion is outside the area of prior radiation; at least 7 days must have elapsed since last radiation treatment; patients must have recovered from any adverse events from prior radiation therapy to =< CTCAE grade 1
* PRIOR/CONCURRENT THERAPY CRITERIA: Patients must not have had a major surgery within 28 days prior to registration; patients must have recovered from any adverse effects of prior surgery to the satisfaction of the treating physician; biopsies and central IV access placement are not considered major surgery
* PRIOR/CONCURRENT THERAPY CRITERIA: Because the composition, pharmacokinetics (PK), and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including but not limited to St. John's wort, kava, ephedra [ma huang], ginko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* CLINICAL/LABORATORY CRITERIA: Patients must have Zubrod performance status of 0-2
* CLINICAL/LABORATORY CRITERIA: Absolute neutrophil count (ANC) >= 1500/mcL; these results must be obtained within 28 days prior to registration
* CLINICAL/LABORATORY CRITERIA: Platelet count >= 100,000/mcL; these results must be obtained within 28 days prior to registration
* CLINICAL/LABORATORY CRITERIA: Hemoglobin >= 9 grams/dl; these results must be obtained within 28 days prior to registration
* CLINICAL/LABORATORY CRITERIA: Total bilirubin =< 1.5 x institutional upper limit of normal (IULN); these results must be obtained within 28 days prior to registration
* CLINICAL/LABORATORY CRITERIA: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x IULN (or =< 5 x IULN for patients with known liver metastases); these results must be obtained within 28 days prior to registration
* CLINICAL/LABORATORY CRITERIA: Serum creatinine =< 1.5 x IULN OR measured or calculated creatinine clearance >= 40 mL/min; this result must have been obtained within 28 days prior to registration
* CLINICAL/LABORATORY CRITERIA: Patients must be able to swallow oral medications and must not have a gastro-intestinal disorder with diarrhea as a major symptom or that may alter absorption such as malabsorption syndromes or gastric resection
* CLINICAL/LABORATORY CRITERIA: Patient must not have prior history of interstitial lung disease or pneumonitis
* CLINICAL/LABORATORY CRITERIA: Patients must not have history of significant co-morbid illness inclusive of but not restricted to New York Heart Association class II, congestive cardiac failure, uncontrolled hypertension, history of myocardial infarction, unstable angina, coronary angioplasty, stenting or cerebrovascular accident within 6 months prior to registration or any other illness that in the assessment of the treating physician would compromise the ability of the patient to participate in this study
* CLINICAL/LABORATORY CRITERIA: Patients must have corrected QT (QTc) interval =< 480 msec (using the Bazett's formula) on electrocardiogram (ECG) performed within 42 days prior to registration; history or evidence of current clinically significant uncontrolled arrhythmias are not eligible; however, patients with controlled atrial fibrillation for > 30 days prior to randomization are eligible; patients must not have atrial fibrillation > grade 2 on the screening ECG; patients with CTCAE grade 1-2 atrial fibrillation on their screening ECG must have a second ECG performed prior to registration and more than 30 days from the screening ECG (either before or after) with the most recent ECG showing stable or improving grade of atrial fibrillation
* CLINICAL/LABORATORY CRITERIA: Patients must have a left ventricular ejection fraction (LVEF) >= institutional lower limit of normal (ILLN) by echocardiography (ECHO) or multi-gated acquisition scan (MUGA) within 42 days prior to registration
* CLINICAL/LABORATORY CRITERIA: Patients must not have untreated or unresolved retinopathy or have a history (or current evidence) of retinal vein occlusion determined by an ophthalmology exam within 42 days prior to registration
* CLINICAL/LABORATORY CRITERIA: Patients must not have an immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, or excipients, or to dimethyl sulfoxide (DMSO) or other agents used in the study
* CLINICAL/LABORATORY CRITERIA: Patients must not have a known history of active hepatitis B or C infection (defined as presence of hepatitis [Hep] B surface antigen [sAg] and/or Hep B deoxyribonucleic acid [DNA] and/or Hep C ribonucleic acid [RNA]); patients must not have a known history of human immunodeficiency virus (HIV) seropositivity
* CLINICAL/LABORATORY CRITERIA: No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years; patients with localized prostate cancer who are being followed by an active surveillance program are also eligible
* CLINICAL/LABORATORY CRITERIA: Patients must not be pregnant or nursing due to the risk of fetal or nursing infant harm; women/men of reproductive potential must have agreed to use an effective contraceptive method (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation and for 4 months after the last dose of the drug; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* SPECIMEN SUBMISSION CRITERIA: Patients must be offered optional participation in banking of specimens for future research
* REGULATORY CRITERIA: Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* REGULATORY CRITERIA: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M Gadgeel, Principal Investigator — SWOG Cancer Research Network
Locations (599):
- United States (599):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Middlesex Hospital, Middletown, Connecticut
  - Low Country Cancer Care, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - UChicago Medicine AdventHealth Cancer Institute Hinsdale, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Garnet Health Medical Center, Middletown, New York
  - University of Rochester, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - WG Hefner VA Medical Center, Salisbury, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Integrity Oncology PLLC-Collierville, Collierville, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Gadgeel SM, Miao J, Riess JW, Moon J, Mack PC, Gerstner GJ, Burns TF, Taj A, Akerley WL, Dragnev KH, Laudi N, Redman MW, Gray JE, Gandara DR, Kelly K. Phase II Study of Docetaxel and Trametinib in Patients with KRAS Mutation Positive Recurrent Non-Small Cell Lung Cancer (NSCLC; SWOG S1507, NCT-02642042). Clin Cancer Res. 2023 Sep 15;29(18):3641-3649. doi: 10.1158/1078-0432.CCR-22-3947. PMID 37233987

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 participants were enrolled. However, 4 were found to be ineligible and 2 did not receive protocol treatment and so were not analyzable. Thus only 54 were included in the analysis.
Groups:
- Treatment (Trametinib, Docetaxel): Participants receive trametinib PO on days 1-21. Participants also receive docetaxel IV on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Docetaxel: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Trametinib: Given PO
Period: Overall Study
Arm/Group | Treatment (Trametinib, Docetaxel)
Started | 54
Completed | 0
Not Completed | 54
Not completed — Adverse Event | 22
Not completed — Refusal Unrelated to Adverse Event | 1
Not completed — Progression/Relapse | 28
Not completed — Death | 1
Not completed — Not Protocol Specified | 2

BASELINE CHARACTERISTICS:
Population: Eligible and analyzable participants
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] — Population: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  years
    All Participants | 65 [47 to 78]
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation | 66 [47 to 78]
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation | 63 [48 to 77]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  Participants
    All Participants: Female | 31
    All Participants: Male | 23
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation: Female | 11
    Participants with G12C Mutation: Male | 8
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation: Female | 20
    Participants with Non-G12C Mutation: Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 46
  More than one race | 0
  Unknown or Not Reported | 1
Smoking Status [Count of Participants; unit: Participants] — Population: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  Participants
    All Participants: Current | 12
    All Participants: Former | 38
    All Participants: Never | 4
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation: Current | 2
    Participants with G12C Mutation: Former | 15
    Participants with G12C Mutation: Never | 2
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation: Current | 10
    Participants with Non-G12C Mutation: Former | 23
    Participants with Non-G12C Mutation: Never | 2
Zubrod Performance Status [Count of Participants; unit: Participants] — Participants are graded according to the Zubrod Performance Status Scale, which runs from 0 to 5, with 0 denoting perfect health and 5 death
  0 - fully active, able to carryout pre-disease performance without restriction
  1. - restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework or office work
  2. - ambulatory and capable of self-care but unable to carry out work activities; up and about more than 50% of waking hours Population: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  Participants
    All Participants: 0 | 16
    All Participants: 1 | 37
    All Participants: 2 | 1
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation: 0 | 6
    Participants with G12C Mutation: 1 | 12
    Participants with G12C Mutation: 2 | 1
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation: 0 | 10
    Participants with Non-G12C Mutation: 1 | 25
    Participants with Non-G12C Mutation: 2 | 0
Histology [Count of Participants; unit: Participants] — Population: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  Participants
    All Participants: Adenocarcinoma | 48
    All Participants: Other | 6
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation: Adenocarcinoma | 17
    Participants with G12C Mutation: Other | 2
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation: Adenocarcinoma | 31
    Participants with Non-G12C Mutation: Other | 4
Metastic Sites at Baseline (Liver) [Count of Participants; unit: Participants] — Population: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  Participants
    All Participants | 17
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation | 8
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation | 9
Metastic Sites at Baseline (Brain) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  Participants
    All Participants | 7
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation | 4
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation | 3
Prior Regimens [Count of Participants; unit: Participants] — Population: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  Participants
    All Participants: 1 | 16
    All Participants: 2 | 38
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation: 1 | 6
    Participants with G12C Mutation: 2 | 13
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation: 1 | 10
    Participants with Non-G12C Mutation: 2 | 25
Prior Immunotherapy [Count of Participants; unit: Participants] — Population: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  Participants
    All Participants: Yes | 31
    All Participants: No | 23
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation: Yes | 12
    Participants with G12C Mutation: No | 7
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation: Yes | 19
    Participants with Non-G12C Mutation: No | 16
KRAS Mutation Type [Count of Participants; unit: Participants] — Population: Eligible and analyzable participants were stratified based on whether they had G12C mutation or non-G12C mutations. Baseline measures are reported in separate rows for all participants (54), participants with G12C mutation (19), and participants with non-G12C mutations (35).
  Participants
    All Participants: G12A | 9
    All Participants: G12C | 19
    All Participants: G12D | 9
    All Participants: G12F | 1
    All Participants: G12S | 2
    All Participants: G12V | 7
    All Participants: G13C | 4
    All Participants: G13D | 1
    All Participants: Q61K | 1
    All Participants: Q61L | 1
    Participants with G12C Mutation: number analyzed (Participants) | 19
    Participants with G12C Mutation: G12A | 0
    Participants with G12C Mutation: G12C | 19
    Participants with G12C Mutation: G12D | 0
    Participants with G12C Mutation: G12F | 0
    Participants with G12C Mutation: G12S | 0
    Participants with G12C Mutation: G12V | 0
    Participants with G12C Mutation: G13C | 0
    Participants with G12C Mutation: G13D | 0
    Participants with G12C Mutation: Q61K | 0
    Participants with G12C Mutation: Q61L | 0
    Participants with Non-G12C Mutation: number analyzed (Participants) | 35
    Participants with Non-G12C Mutation: G12A | 9
    Participants with Non-G12C Mutation: G12C | 0
    Participants with Non-G12C Mutation: G12D | 9
    Participants with Non-G12C Mutation: G12F | 1
    Participants with Non-G12C Mutation: G12S | 2
    Participants with Non-G12C Mutation: G12V | 7
    Participants with Non-G12C Mutation: G13C | 4
    Participants with Non-G12C Mutation: G13D | 1
    Participants with Non-G12C Mutation: Q61K | 1
    Participants with Non-G12C Mutation: Q61L | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Confirmed and Unconfirmed Complete and Partial Responses) in All KRAS Mutant Participants
Description: Proportion of participants who have a partial or complete response to treatment per RECIST v1.1
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 3 years
Population: All eligible and analyzable participants
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 54
proportion of participants | 0.33 [0.21 to 0.47]

2. Secondary Outcome: Response Rate (Confirmed and Unconfirmed Complete and Partial Responses) in Participants With G12C KRAS Mutation
Description: as for outcome 1
Time Frame: Up to 3 years
Population: Eligible and analyzable participants with G12C KRAS mutation
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 19
proportion of participants | 0.26 [0.09 to 0.51]

3. Secondary Outcome: Response Rate (Confirmed and Unconfirmed Complete and Partial Responses) in Participants With Non-G12C KRAS Mutation
Description: as for outcome 1
Time Frame: up to 3 years
Population: Eligible and analyzable participants with Non-G12C mutation
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 35
proportion of participants | 0.37 [0.21 to 0.55]

4. Secondary Outcome: Progression Free Survival in All KRAS Mutant Participants
Description: Time from date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed using the same techniques as baseline, as well as absolute increase of at least 0.5 cm; unequivocal progression of non-measurable disease; appearance of any new lesion/site; death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: Up to 3 years
Population: All eligible and analyzable participants
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 54
months | 4.1 [3.1 to 5.1]

5. Secondary Outcome: Progression Free Survival in Participants With G12C KRAS Mutation
Description: Time from date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed using the same techniques as baseline, as well as absolute increase of at least 0.5 cm; unequivocal progression of non-measurable disease; appearance of any new lesion/site; death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: Up to 3 years
Population: Eligible and analyzable participants with G12C KRAS mutation
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 19
months | 3.3 [1.5 to 4.3]

6. Secondary Outcome: Progression Free Survival in Participants With Non-G12C KRAS Mutation
Description: as for outcome 5
Time Frame: Up to 3 years
Population: Eligible and analyzable participants with non-G12C KRAS mutation
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 35
months | 4.1 [3.4 to 5.6]

7. Secondary Outcome: Overall Survival in All KRAS Mutants
Description: Time from date of registration to date of death due to any cause.
Time Frame: Up to 3 years
Population: All eligible and analyzable participants
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 54
months | 10.9 [8.0 to 14.0]

8. Secondary Outcome: Overall Survival in Participants With G12C KRAS Mutation
Description: Time from date of registration to date of death due to any cause.
Time Frame: Up to 3 years
Population: Eligible and analyzable participants with G12C KRAS mutation
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 19
months | 8.8 [4.9 to 10.9]

9. Secondary Outcome: Overall Survival in Participants With Non-G12C KRAS Mutation
Description: Time from date of registration to date of death due to any cause.
Time Frame: up to 3 years
Population: Eligible and analyzable participants with non-G12C KRAS mutation
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 35
months | 12.2 [8.0 to 18.8]

10. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Patients who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Treatment (Trametinib, Docetaxel)
Number analyzed (Participants) | 54
Participants
  Abdominal pain | 1
  Alanine aminotransferase increased | 1
  Anemia | 4
  Anorexia | 2
  Aspartate aminotransferase increased | 2
  Colitis | 1
  Conjunctivitis | 1
  Dehydration | 2
  Diarrhea | 5
  Dyspnea | 4
  Ejection fraction decreased | 1
  Electrocardiogram QT corrected interval prolonged | 1
  Fatigue | 8
  Febrile neutropenia | 2
  Gastrointestinal disorders - Other, specify | 2
  Generalized muscle weakness | 1
  Hyperkalemia | 2
  Hypermagnesemia | 1
  Hypokalemia | 2
  Hyponatremia | 3
  Hypotension | 2
  Hypoxia | 1
  Left ventricular systolic dysfunction | 1
  Lung infection | 5
  Lymphocyte count decreased | 1
  Mucositis oral | 4
  Multi-organ failure | 1
  Myocardial infarction | 1
  Nausea | 3
  Neutrophil count decreased | 4
  Palmar-plantar erythrodysesthesia syndrome | 1
  Pericardial effusion | 1
  Peripheral sensory neuropathy | 1
  Pneumonitis | 2
  Pruritus | 2
  Rash acneiform | 3
  Rash maculo-papular | 8
  Rash pustular | 1
  Respiratory failure | 2
  Restrictive cardiomyopathy | 1
  Sepsis | 6
  Stroke | 1
  Thromboembolic event | 2
  Upper gastrointestinal hemorrhage | 1
  Urinary tract infection | 1
  Vomiting | 2
  White blood cell decreased | 2
  Wound infection | 1

11. Other Pre Specified Outcome: Response Rates in the Presence of p53 Mutations
Description: The response rate between patients with dysfunctional p53 will be compared to the response rate in patients without p53 dysfunction.
Time Frame: Up to 3 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Response Rates in the Presence of LKB1 Mutations
Description: The response rate between patients with LKB1 disruption will be compared to the response rate in patients without LKB1 disruption. The response rate will be estimated by LKB1 disruption status (yes/no), along with 95% confidence intervals around the estimated proportions. This analysis will evaluate if disruption in LKB1 is associated with a lower probability of response.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Description: 54 participants who were eligible and received protocol therapy were assessed for AEs.
Arm/Group | Treatment (Trametinib, Docetaxel)
All-Cause Mortality (participants affected / at risk) | 44/54
Serious Adverse Events (participants affected / at risk) | 31/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib, Docetaxel) (N=54)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Lung infection (Infections and infestations) | 7
Sepsis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Stroke (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trametinib, Docetaxel) (N=54)
Anemia (Blood and lymphatic system disorders) | 27
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders-Other (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 7
Ventricular arrhythmia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 5
Conjunctivitis (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Eye disorders-Other (Eye disorders) | 4
Glaucoma (Eye disorders) | 1
Watering eyes (Eye disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 13
Anal pain (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 22
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 39
Dry mouth (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 32
Oral hemorrhage (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 16
Chills (General disorders) | 4
Edema face (General disorders) | 3
Edema limbs (General disorders) | 19
Fatigue (General disorders) | 44
Fever (General disorders) | 12
Flu like symptoms (General disorders) | 1
General disorders and admin site conditions - Other (General disorders) | 4
Infusion related reaction (General disorders) | 1
Malaise (General disorders) | 1
Multi-organ failure (General disorders) | 1
Neck edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 2
Bronchial infection (Infections and infestations) | 1
Infections and infestations-Other (Infections and infestations) | 4
Laryngitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 4
Papulopustular rash (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Periorbital infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 2
Sepsis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 4
Upper respiratory infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 3
Vaginal infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 15
Aspartate aminotransferase increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 2
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 6
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
INR increased (Investigations) | 1
Investigations-Other (Investigations) | 4
Lymphocyte count decreased (Investigations) | 10
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 9
Weight gain (Investigations) | 3
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 10
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 11
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 24
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 18
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Ataxia (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 8
Dysphasia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Lethargy (Nervous system disorders) | 1
Nervous system disorders-Other (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 7
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 2
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 5
Acute kidney injury (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Renal and urinary disorders-Other (Renal and urinary disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 17
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 4
Nail loss (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash acneiform (Skin and subcutaneous tissue disorders) | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 9
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 2
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 15
Hypotension (Vascular disorders) | 8
Thromboembolic event (Vascular disorders) | 3
Vascular disorders-Other (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT02642042/Prot_SAP_000.pdf